CLINICAL TRIAL: NCT01144949
Title: A Double-Blind, Placebo-Controlled Study of Silodosin to Facilitate Urinary Stone Passage
Brief Title: Study of Silodosin to Facilitate Passage of Urinary Stones
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIL1001
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Ureteral Calculi; Kidney Stones; Urolithiasis
Keywords: ureteral calculi; renal colic; ureteral stones; kidney stones; medical expulsive therapy
MeSH Terms: conditions — Ureteral Calculi; Kidney Calculi; Urolithiasis; Renal Colic | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- silodsosin (Active Comparator)
  Interventions: Drug: silodosin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: silodosin — one silodosin 8 mg capsule orally, once daily, with food for up to 4 weeks
  Arms: silodsosin
Drug: placebo — one placebo capsule orally, once daily, with food for up to 4 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to assess if patients treated with silodosin will have a higher spontaneous passage rate of their ureteral stone than those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older
* Male or a non-pregnant, non-lactating female using adequate means of birth control, if not menopausal
* Have radiopaque unilateral ureteral calculus ≥4mm and ≤10mm in any location of the ureter

Exclusion Criteria:

* Multiple ureteral calculi, or a solitary kidney, or refractory renal colic, or a non-opaque calculus, or active urinary tract infection, or severe hydronephrosis
* History of previous ureteral surgery or ureteral stricture on affected side
* History of any of the following conditions: myasthenia gravis, myopathy, spina bifida, spinal cord injury, autonomic nervous system disorder, fibromyalgia, breast cancer
* Moderate to severe renal impairment or severe liver insufficiency
* History of significant postural hypotension
* Is receiving medication(s) which preclude safe participation in the study or that may produce a confounding effect on the variables under study
* History of allergy to alpha-blockers or oxycodone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Olsen, MPH, Study Director — Watson Pharmaceuticals, Inc.
Locations (27):
- United States (27):
  - Watson Investigational Site, Birmingham, Alabama
  - Watson Investigational Site, Anchorage, Alaska
  - Watson Investigative Site, Mission Hills, California
  - Watson Investigational Site, Murrieta, California
  - Watson Investigational Site, San Diego, California
  - Watson Investigational Site, Daytona Beach, Florida
  - Watson Investigational Site, Gainesville, Florida
  - Watson Investigational Site, Orange City, Florida
  - Watson Investigative Site, Overland Park, Kansas
  - Watson Investigative Site, North Kansas City, Missouri
  - Watson Investigational Site, Hackensack, New Jersey
  - Watson Investigational Site, Mount Laurel, New Jersey
  - Watson Investigational Site, Sewell, New Jersey
  - Watson Investigational Site, Voorhees Township, New Jersey
  - Watson Investigational Site, Albany, New York
  - Watson Investigational Site, Garden City, New York
  - Watson Investigational Site, New York, New York
  - Watson Investigational Site, Plainview, New York
  - Watson Investigational Site, Syracuse, New York
  - Watson Investigational Site, Cincinnati, Ohio
  - Watson Investigational Site, Columbus, Ohio
  - Watson Investigational Site, Bala-Cynwyd, Pennsylvania
  - Watson Investigational Site, Lancaster, Pennsylvania
  - Watson Investigational Site, Myrtle Beach, South Carolina
  - Watson Investigational Site, Dallas, Texas
  - Watson Investigational Site, San Antonio, Texas
  - Watson Investigational Site, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silodsosin | Placebo
Started | 119 | 120
Completed | 108 | 106
Not Completed | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silodsosin | Placebo | Total
Number analyzed (Participants) | 119 | 120 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.5) | 46.7 (15.2) | 47.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 36 | 83
  Male | 72 | 84 | 156

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Stone Passage (Distal Stones) Without Need for Emergency Department Visits, Hospital Admissions, Surgical Intervention, or Other Interventional Procedures.
Description: The primary efficacy variable is the occurrence of spontaneous distal stone passage within 4 weeks, as determined by radiography.
  For this outcome measure, analysis includes only those stones located in the distal ureter.
Time Frame: 4 weeks
Population: Those subjects in the ITT population (defined as randomized and received at least one dose of study drug) with stones located in the distal ureter (determined by radiography) were included in this analysis. The number of ITT subjects with distal stones was 52/115 in the 8 mg silodosin treatment arm and 59/117 in the placebo treatment arm.
Measure: Number; unit: participants
Arm/Group | Silodsosin | Placebo
Number analyzed (Participants) | 52 | 59
participants | 36 | 27

2. Secondary Outcome: Time to Spontaneous Stone Passage (Distal Stones)
Description: Time to stone passage for distally-located stones is assessed by entries in subject diaries.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Silodsosin | Placebo
Number analyzed (Participants) | 52 | 59
days | 19.6 (1.61) [12 to 29] | 22.0 (1.47) [lower limit 26]

3. Secondary Outcome: Outpatient Narcotic Analgesic Use for Pain Relief
Description: Narcotic analgesic use was assessed through a subject diary. Analysis was performed on the number of days with analgesic use.
Time Frame: 4 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Silodsosin | Placebo
Number analyzed (Participants) | 95 | 104
Days | 5.8 (8.0) | 5.5 (6.8)

4. Secondary Outcome: Change From Baseline in Average Score on the Brief Pain Inventory (Distal Stones)
Description: At each study visit, subjects were given a Brief Pain Inventory (BPI) Questionnaire to complete. The BPI collects subject-reported pain severity scores and assesses impact of pain upon the subject's daily life, on a 10-point scale (with 10 being the greatest severity/impact). Analysis was change from baseline to week 4.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silodsosin | Placebo
Number analyzed (Participants) | 52 | 59
units on a scale | -2.6 (2.5) | -1.9 (3.1)

5. Primary Outcome: Spontaneous Stone Passage (All Stones) Without Need for Emergency Department Visits, Hospital Admissions, Surgical Intervention, or Other Interventional Procedures.
Description: The primary efficacy variable is the occurrence of spontaneous stone passage within 4 weeks, as determined by radiography. For this outcome measure, analysis includes all ureteral stones, regardless of location in the ureter.
Time Frame: 4 weeks
Population: This endpoint analyzed all subjects in the ITT population, defined as randomized and received at least one dose of study drug (115 in the 8 mg silodosin arm, 117 in the placebo arm)
Measure: Number; unit: participants
Arm/Group | Silodsosin | Placebo
Number analyzed (Participants) | 115 | 117
participants | 60 | 52

6. Secondary Outcome: Time to Spontaneous Stone Passage (All Stones)
Description: Time to stone passage for all ureteral stones (regardless of location) is assessed by entries in subject diaries.
Time Frame: 4 weeks
Population: ITT population
Measure: Mean (Standard Error); unit: days
Arm/Group | Silodsosin | Placebo
Number analyzed (Participants) | 115 | 117
days | 22.3 (1.02) [26 to 31] | 22.9 (1.00) [lower limit 26]

ADVERSE EVENTS:
Arm/Group | Silodsosin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/119 | 2/120
Other Adverse Events (participants affected / at risk) | 27/119 | 8/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silodsosin (N=119) | Placebo (N=120)
Renal colic (Renal and urinary disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Silodsosin (N=119) | Placebo (N=120)
Retrograde ejaculation (Reproductive system and breast disorders) | 11 | 1
Nausea (Gastrointestinal disorders) | 9 | 2
Dizziness (Nervous system disorders) | 8 | 2
Headache (Nervous system disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less